CLINICAL TRIAL: NCT04943003
Title: Neurobiological Predictors of Response to Non-invasive Neurostimulation and Genetic Susceptibility to Dementia in Patients With Amnestic Mild Cognitive Impairment (CCL)
Brief Title: Study of Neurobiological Predictors of Response to Non-invasive Neurostimulation and Genetic Susceptibility to Dementia in Patients With Amnestic Mild Cognitive Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Suellen Marinho Andrade (Other)
Responsible Party: Sponsor-Investigator, Suellen Marinho Andrade, Principal Investigator, Federal University of Paraíba
Organization: Federal University of Paraíba (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS in MCI
Record Dates: First submitted 2021-06-06; First posted 2021-06-29 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; tDCS; Computational modeling
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be divided into 02 groups, each with 25 patients, totaling 50 volunteers: Active - participants who will receive real current; Sham - participants who will receive simulated stimulation. Participants entered into the study through the eligibility criteria will be randomly allocated in a simple way, at a rate of 1:1.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All examiners will be blinded to the type of treatment the patient received (active stimulation or sham) and other assessments. Thus, all guidelines established by CONSORT 2010 (Consolidated Standards of Reporting Trials) will be complied with, as pointed out by Moher et al. (2010), with variable control following systematized and countersigned procedures: random sequence generation, allocation concealment, blinding of participants and professionals, blinding of outcome evaluators and attrition bias (loss analysis using the last observation carried forward method) (Higgins & Green, 2011).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): SimNIBS will be used for modeling. It is a free and open source software package for the simulation of electric field induced by tDCS in the individual brain.
  Modeling will be done using T1-weighted anatomical images of each subject to reconstruct a high-resolution head model of each individual. For electrode placement, we will simulate areas F5 and F6, according to the EEG 10-20 system, for the anode and cathode, respectively, targeting the left and right Dorsolateral Prefrontal Cortex (DLPFC). This group will receive active tDCS, for 30 minutes and for 5 consecutive days, in two weeks, with an anode positioned on the left DLPFC and a cathode electrode placed on the right supraorbital area.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS (Sham Comparator): The electrodes will be placed in the same way as in the Active tDCS group. However, individuals in this group will receive a stimulation that will last only 20-30 seconds. Afterwards, the device will be turned off, no longer emitting current.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — Initially, a measuring tape will be used to make the markings and measurements necessary for placing the electrodes.
  Regarding neurostimulation, the tDCS device is simple and portable, consisting of four main components: two electrodes (anode and cathode), an ammeter (electric current intensity meter), a potentiometer (voltage controller between electrodes) and a set of batteries. We will use the TCT-Research Neurostimulator, developed by Trans Cranial Technologies (Hong Kong, China), Regarding the protocols, the Active tDCS group will receive active tDCS for 30 minutes and for 5 consecutive days, in two weeks, with an anode positioned on the left DLPFC and a cathode electrode placed on the right supraorbital area. The 10-20 International EEG system will be taken as a reference. The current intensity will be defined from computational modeling, using Nuclear Magnetic Resonance (NMR) to estimate and individualize the dose to be administered.

SUMMARY:
Transcranial Direct Current Stimulation is a non-invasive neuromodulatory technique that results in the clinical improvement of patients with Mild Cognitive Impairment, a prodromal condition for the onset of dementia. The responses to treatment depend on the characteristics of the patients and the parameters adjusted in the equipment, which makes the modeling of electric fields imperative to maximize the safety profile and therapeutic potential of the technique. The study of neurobiological predictors of response to non-invasive neurostimulation and genetic susceptibility can elucidate current effects according to the individual's profile. The objectives of this study are to observe the effects of Transcranial Direct Current Stimulation with optimized/customized parameters in patients with amnestic CCL, considering the subjects' genetic susceptibility to Alzheimer's Disease and neurobiological markers. This is a randomized, triple-blind, sham-controlled clinical trial. Neuropsychological tests and a sociodemographic and clinical questionnaire will be used to assess and characterize the subjects. Participants captured by the Laboratory of Studies in Aging and Neuroscience at the Federal University of Paraíba will be divided into 02 groups, each with 25 patients, totaling 50 volunteers: Active - participants who will receive real current; Sham - participants who will receive simulated stimulation. Participants entered through the eligibility criteria will be randomly allocated in a simple way, at a rate of 1:1. Payment parameters will be customized by Computational Modeling with the aid of the SimNIBS Program and Nuclear Magnetic Resonance. The electroencephalogram and evaluation of polymorphisms of the gene encoding Apolipoprotein E examined as predictors of response. Data will be processed from the Statistical Package for Social Sciences® (20.0) Software, applying the Student test for continuous variables or chi-square for categorical variables. Predictive analysis will be conducted from Machine Learning. It is expected to find improvements in the scores of memory and general cognition tests after the intervention protocol with tDCS with individualized dose in the group that will receive an intervention, compared to the simulated neurostimulation group. These obtained results optimize the practice, elucidating issues still present due to the different applications of the technique produced in the literature on the subject.

DETAILED DESCRIPTION:
Neuropsychological tests and a sociodemographic and clinical questionnaire will be used to assess and characterize the subjects. Participants captured by the Laboratory of Studies in Aging and Neuroscience at the Federal University of Paraíba will be divided into 02 groups, each with 25 patients, totaling 50 volunteers: Active - participants who will receive real current; Sham - participants who will receive simulated stimulation. Participants entered through the eligibility criteria will be randomly allocated in a simple way, at a rate of 1:1. Payment parameters will be customized by Computational Modeling with the aid of the SimNIBS Program and Nuclear Magnetic Resonance. The electroencephalogram and evaluation of polymorphisms of the gene encoding Apolipoprotein E examined as predictors of response.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with Mild Cognitive Impairment (MCI);
* Both sexes;
* Aged 65 years or older, without a diagnosis of dementia will be included.

Exclusion Criteria:

* Unstable medical conditions;
* Patients with metallic implants and pacemakers;
* Epileptics;
* Using drugs/alcohol, regular use of hypnotics and benzodiazepines up to two weeks before the start of the study;
* People who have been using medication with cholinergic inhibitors for more than two months before this clinical trial

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-26 (Estimated); Primary Completion 2022-12-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Examination (MMSE) (T0) | The evoluations will be carried out in Pre-intervention (T0)
  To assess the primary outcome, the Mini Mental State Examination (MMSE) o will be used, developed in the United States and published in 1975, whose maximum score is 30 points and includes questions about memory, attention , orientation, language, and visuospatial skills.
  We will adopt the 24-point score for the standard cut, following recommendations expressed in the literature. In order to avoid false positives and false negatives, we will perform the stratification by levels or years of schooling, as educational level is the main predictor of MMSE performance.
  Authors recorded good internal consistency (0.62 to 0.79) and a high test-retest reliability of the MMSE, ranging from 0.76 to 0.90, being a reliable instrument to detect CCL and AD .
Mini Mental State Examination (MMSE) (T1) | The evoluations will be performed up to one week after the stimulation protocol (T1)
  To assess the primary outcome, the Mini Mental State Examination (MMSE) o will be used, developed in the United States and published in 1975, whose maximum score is 30 points and includes questions about memory, attention , orientation, language, and visuospatial skills.
  We will adopt the 24-point score for the standard cut, following recommendations expressed in the literature. In order to avoid false positives and false negatives, we will perform the stratification by levels or years of schooling, as educational level is the main predictor of MMSE performance.
  Authors recorded good internal consistency (0.62 to 0.79) and a high test-retest reliability of the MMSE, ranging from 0.76 to 0.90, being a reliable instrument to detect CCL and AD .

SECONDARY OUTCOMES:
Digit Span Memory Test | The evoluations will be carried out in Pre-intervention (T0)
  This is one of the main tasks used in short-term memory assessment, where the examiner asks the patient to repeat a series of numbers (eg 2-5, 3-6-7). The first sequence starts with two digits, and after each correct answer the examiner adds one digit to the next sequence. The test is composed of two parts, in forward and reverse order, allowing the assessment of short-term memory storage capacity and its executive component.
Digit Span Memory Test | The evoluations will be performed up to one week after the stimulation protocol (T1)
  This is one of the main tasks used in short-term memory assessment, where the examiner asks the patient to repeat a series of numbers (eg 2-5, 3-6-7). The first sequence starts with two digits, and after each correct answer the examiner adds one digit to the next sequence. The test is composed of two parts, in forward and reverse order, allowing the assessment of short-term memory storage capacity and its executive component.
Beck Depression Scale II and Beck Anxiety Inventory | The evoluations will be carried out in Pre-intervention (T0)
  The Beck II Depression Scale, a self-report instrument for depression, has 21 items that reveal how the individual has felt during the last two weeks (including the current day), in which there are four answers for each one (with a score ranging from 0 to 3). The total score is the sum of individual items, whose maximum score can reach 63 points, being classified into levels: mild, moderate and severe.
  The Beck Anxiety Inventory consists of 21 items that assess how the individual has been feeling during the last two weeks, including the current day, enabling the collection of information about anxiety symptoms. Each item has 4 options, among which one can be chosen by the participant (ranging from 0 to 3 the score of each option). The total score is calculated by adding the individual response for each item, with a maximum score of 63 points. The results will be used as a prediction of response to neurostimulation.
Beck Depression Scale II and Beck Anxiety Inventory | The evoluations will be performed up to one week after the stimulation protocol (T1)
  The Beck II Depression Scale, a self-report instrument for depression, has 21 items that reveal how the individual has felt during the last two weeks (including the current day), in which there are four answers for each one (with a score ranging from 0 to 3). The total score is the sum of individual items, whose maximum score can reach 63 points, being classified into levels: mild, moderate and severe.
  The Beck Anxiety Inventory consists of 21 items that assess how the individual has been feeling during the last two weeks, including the current day, enabling the collection of information about anxiety symptoms. Each item has 4 options, among which one can be chosen by the participant (ranging from 0 to 3 the score of each option). The total score is calculated by adding the individual response for each item, with a maximum score of 63 points. The results will be used as a prediction of response to neurostimulation.
Genetic susceptibility (ApoE) | The evoluations will be carried out in Pre-intervention (T0)
  For ApoE allele genotyping, the researchers will follow the recommendations proposed by Crook, Hardy & Duff (1994) and Wenham, Newton, & Price (1991), and the genomic DNA will be amplified by a Polymerase Chain Reaction (PCR). The results will be used as a prediction of response to neurostimulation.
Electroencephalography | The evoluations will be carried out in Pre-intervention (T0)
  Brain electrical activity will be captured using the BrainVision actiCHamp32 equipment (Brain vision, Herrsching, Germany), using 32 Ag/AgCl electrodes, which will be positioned and fixed based on the 10-20 International System. The data will be used to assess brain electrical activity at baseline.
Electroencephalography (EEG) | The evoluations will be performed up to one week after the stimulation protocol (T1)
  Brain electrical activity will be captured using the BrainVision actiCHamp32 equipment (Brain vision, Herrsching, Germany), using 32 Ag/AgCl electrodes, which will be positioned and fixed based on the 10-20 International System. The regions of interest to be monitored are: prefrontal, frontal, parietal, temporal and occipital region, bilaterally (Fz, F3, F7, FT9, FC5, FC1, C3, T7, TP9, CP5, CP1, Pz, P3, P7, O1, Oz, O2, P4, P8, TP10, CP6, CP2, Cz, C4, T8, FT10, FC6, FC2, F4, F8, Fp2, Fp1), in the silent condition in the eyes and eyes closed states , for five minutes each, totaling 10 minutes of collection for each subject. The results will be used as a prediction of response to neurostimulation.
Magnetic Resonance Imaging-MRI | The evoluations will be carried out in Pre-intervention (T0)
  High-resolution anatomical images will be acquired using a T1-weighted fast gradient sequence prepared by three-dimensional magnetization with the following parameters: repetition time (TR) = 1900ms, echo time (TE) = 2.2 ms, inversion time (TI) = 900 ms, inversion angle (FA) = 9°, number of slices = 176, slice thickness = 1 mm, voxel size = 1 × 1 × 1 mm 3 and matrix = 256 × 256. The results will be used for computational modeling and to assess brain electrical activity at baseline.
Magnetic Resonance Imaging-MRI | The evoluations will be performed up to one week after the stimulation protocol (T1)
  High-resolution anatomical images will be acquired using a T1-weighted fast gradient sequence prepared by three-dimensional magnetization with the following parameters: repetition time (TR) = 1900ms, echo time (TE) = 2.2 ms, inversion time (TI) = 900 ms, inversion angle (FA) = 9°, number of slices = 176, slice thickness = 1 mm, voxel size = 1 × 1 × 1 mm 3 and matrix = 256 × 256. The results will be used as a prediction of response to neurostimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Paraíba,Department of Psychology, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No